CLINICAL TRIAL: NCT02870244
Title: Adoptive T Cell Immunotherapy for Advanced Melanoma Using Engineered Lymphocytes: A Phase 1b Study
Brief Title: Adoptive T Cell Immunotherapy for Advanced Melanoma Using Engineered Lymphocytes
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Loyola University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michael Nishimura, Professor, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 203729
Record Dates: First submitted 2016-07-22; First posted 2016-08-17 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Melanoma
Keywords: Melanoma; Gene Therapy; Adoptive T-Cell Transfer; IL-2
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Escalating Doses (Experimental): Three patients will be treated at the first & each subsequent dose level. Patients will be observed for 30 days post T cell infusion. If there was one DLT in the first 3 patients, an additional 3 patients will be treated at that level. If no additional DLTs are observed (for a total of 1 DLT in 6 patients) then the dose will be escalated. If two patients in the first 3 patients at a dose level experience a DLT, the dose will be de-escalated to the previous level & an additional 3 patients will be enrolled at that level if 6 have not yet been treated at that level. The maximum tolerated dose (MTD) is defined as the highest dose at which 0 or 1 patient in six has experienced a DLT. If 2 or 3 patients in the first 3 patients experience a DLT at the first dose level, the study will terminate.
  Interventions: Biological: Escalating Doses

INTERVENTIONS:
Biological: Escalating Doses — Subjects will receive a single infusion of autologous bulk TIL 13831 TCR transduced T cells supported with low dose IL-2. Autologous bulk TIL 13831 TCR transduced T cells means the infusion will consist of a polyclonal mixture of CD4 + and CD8+ T Cells expressing the TIL 13831 TCR.
  Subjects in Cohort 1 will receive 7.5 x 10^6/kg TIL 1383I TCR transduced T cells.
  Subjects in Cohort 2 will receive 2.5 x 10^7/kg TIL 1383I TCR transduced T cells.
  Subjects in Cohort 3 will receive 7.5 x 10^7/kg TIL 1383I TCR transduced T cells.

SUMMARY:
Phase I clinical trial to determine the Phase II dose of autologous TIL 1383I TCR gene modified T Cells using a retrovirus. This is a novel National Cancer Institute (NCI) funded investigator initiated therapy for patients with advanced melanoma.

DETAILED DESCRIPTION:
This is a Phase 1 dose escalation study designed to find the highest dose of TIL 1383I TCR transduced T cells that can safely be given. Three cohorts of 3 patients will be treated with increasing doses of TIL 1383I TCR transduced T cells. Patients will be monitored clinically and immunologically for a year after infusion. Subjects in Cohort 1 will receive 7.5 X 10^6/kg TIL 1383I TCR transduced T cells. Subjects in Cohort 2 will receive 2.5 x 10^7/kg TIL 1383I TCR transduced T cells. Subjects in Cohort 3 will receive 7.5 x 10^7/kg TIL 1383I TCR transduced T cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of metastatic melanoma which is evaluable either clinically or radiologically.
* Patients must be 18 years of age or older.
* Patients must consent to be in the study and must have signed and dated an approved consent form, which conforms to federal and institutional guidelines.
* Patients must have a performance status (PS) of 0 or 1 ECOG PS scale.
* Patients must have the ability to provide written informed consent prior to study specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time.
* Patients melanoma must be positive for both tyrosinase and HLA-A2 pathologic review from FNA, core or excisional biopsy of lesion.
* Cardiac ejection fraction greater than 50 percent as determined by screening echocardiogram.
* Patients that have undergone treatment with anti-CTLA-4, Cytotoxic T-Lymphocyte Antigen 4, antibody must have at least 6 weeks from last dose of CTLA-4 antibody and evidence of tumor progression before they can be enrolled into this study.
* Patients that have undergone treatment with anti-PD-1, Programmed Death Receptor 1, Blockade or anti-PD-L1 antibody must have at least 4 weeks from last dose of antibody and evidence of tumor progression before they can be treated in this study.
* Patients with V600E mutations are eligible if they have failed an approved BRAF inhibitor or MEK inhibitor therapy or have refused treatment with an approved BRAF inhibitor or MEK inhibitor.
* Patients treated with prior Interleukin-2 (IL-2) are eligible.
* Sufficient cardiopulmonary reserve for IL-2 per institutional guidelines.

Exclusion Criteria:

* Special classes of subjects such as fetuses, pregnant women, children, prisoners, institutionalized individuals, or others who are likely to be vulnerable.
* ECOG performance status of 2 or greater.
* Patients with a history metastatic melanoma involving the brain will be excluded if they have active disease or have had active disease within the prior three months that was not controlled with surgery or radiotherapy.
* Patients taking steroids for disease control or pain management
* Patients must not be pregnant or nursing because of the potentially harmful effects of these agents on a developing fetus. Women or men of reproductive potential must have agreed to use an effective contraceptive method.
* Patients whose BRAF V600 mutation status is unknown should undergo an attempt to determine this information, patients who have a BRAF V600 mutation and are responding to BRAF with or without MEK inhibitor therapy, or have a BRAF V600 mutation and have not been offered the option of receiving BRAF with or without MEK inhibitor therapy for the treatment of their melanoma are excluded.
* No prior malignancy is allowed except for the following- adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for two years.
* Patients that have undergone immunotherapy targeting tyrosinase.
* Patients that have undergone immunotherapy in combination with non-myeloablative chemotherapy.
* Any of the following abnormal laboratory values Absolute neutrophil count less than 1.5 x 10^9/L Platelet count less than 100 x 10^9/L Serum bilirubin greater than 1.5 x upper limit of normal ULN Serum ALT, AST greater than 2.5 x ULN Serum ALP greater than 2 x ULN Serum Albumin less than 2.5 g dL International Normalized Ratio, INR greater than 1.5 Serum creatinine calculated creatinine clearance by the method of Cockcroft and Gault, less than 50mL min.
* Patients should not have any evidence of active or uncontrolled infection requiring treatment with antibiotics.
* Any severe or poorly controlled systemic disease, for example hypertension, clinically significant cardiovascular, pulmonary, or metabolic disease, disorders of wound-healing, ulcer or bone fracture.
* Patients who have received any chemotherapy or investigational treatment within 4 weeks of study start.
* Known infection with HIV, HBV, or HCV.
* Known hypersensitivity to any of the components of the study drugs.
* Patients assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2015-02 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Approximately 18 patients with Grade 2 through Grade 5 Adverse Events that are related to study drug, graded according to NCI CTCAE Version 4.0 | 4 weeks
  Establish a recommended phase II dose of autologous T cell receptor transduced T cells by evaluating unexpected Grade 2 adverse events through Grade 5 regardless of attribution, all toxicities attributed to the cells, and all incidences of intubation including the duration and reason for intubation.

SECONDARY OUTCOMES:
Immunologic changes in T cell count | Baseline and 4 weeks
  Change in T cell count from baseline to 4 weeks.
Audiologic changes of Grade 2 or higher as related to study drug, graded according to NCI CTCAE Version 4.0 | Baseline and 4 weeks
  Potential auditory changes from baseline to 4 weeks.
Ophthalmologic changes or development of Uveitis of Grade 2 or higher as related to study drug, graded according to NCI CTCAE Version 4.0 | Baseline and 4 weeks
  Potential visual changes from baseline to 4 weeks.
CT scans or physical examination from approximately 18 patients will be used to evaluate for a clinical objective response using RECIST Guideline Version 1.1 | Baseline and 4 weeks
  CT scan or physical examination will be used to evaluate for a clinical objective response in patients who have received transduced T Cells at scheduled time points.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Nishimura, PhD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided